CLINICAL TRIAL: NCT01495715
Title: Study With Idebenone in Patients With Chronic Vision Loss Due to Leber's Hereditary Optic Neuropathy (LHON)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNT-III-011
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Leber's Hereditary Optic Neuropathy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — idebenone

ARMS (2):
- Idebenone (Experimental)
  Interventions: Drug: Idebenone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Idebenone
  Arms: Idebenone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to determine whether administration of idebenone can shorten the time to improvement of visual acuity in patients with chronic vision loss due to LHON.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal 10 years and < 65 years
* Impaired visual acuity in affected eyes due to LHON: Visual acuity in best eye >0.4 logMAR
* No explanation for visual loss besides LHON

Exclusion Criteria:

* Any previous use of idebenone
* Participation in another clinical trial of any investigational drug within 3 months prior to Baseline
* Previous participation in Study SNT-II-003 (RHODOS) for idebenone.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)